CLINICAL TRIAL: NCT05066737
Title: Evaluation of the Results of Lateral Suspension Surgeries Performed With the V-NOTES (Vaginal-Natural Orifice Transluminal Endoscopic Surgery) Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Süleyman Salman, associate professor, Gaziosmanpasa Research and Education Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREHf
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; lateral suspension; v-notes; pop-q; pısq-12
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients who has pelvic organ prolapse and underwent lateral suspension via V-notes surgery (Experimental)
  Interventions: Procedure: lateral suspension via V-NOTES surgery

INTERVENTIONS:
Procedure: lateral suspension via V-NOTES surgery — pop-q, pisq-12 assesment of patients with pelvic organ prolapse before and 6 or 12 month after lateral suspension surgery performed via V-NOTES technique.

SUMMARY:
It was aimed to evaluate the quality of life and sexual function of patients by Pre- and postoperative POP-Q (Pelvic Organ Prolapse Quantification) staging and PISQ-12 (Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire) test of patients who underwent lateral suspension operation with V-NOTES (Vaginal-Natural Orifice Transluminal Endoscopic Surgery) Technique.

DETAILED DESCRIPTION:
NOTES technically means a surgical intervention performed by entering the abdomen through one of the body's natural openings such as mouth, anus, vagina, and urethra. With the flexible endoscope, a hole is made in organs such as stomach, colon, vagina, bladder, and the peritoneal cavity is entered and the area to be studied is provided by filling air. With the V-NOTES (vaginal Vaginal-Natural Orifice Transluminal Endoscopic Surgery) method we will apply, we reject the bladder from the cervix and reach to abdominal cavity by piercing the visceral peritoneum. The abdomen will be viewed via trocars placed in this region and a lateral suspension operation, which is a kind of suspension surgery of pelvic organ prolapsus, will be performed.The POP-Q staging that will be performed before the lateral suspension operation with the V-NOTES Technique will be compared with the POP-Q staging 6 after the operation. In addition, Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) test will be used for the evaluation of pelvic organ prolapse, urinary incontinence and sexual function in the same intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 2nd and 3rd degree uterine prolapsus
* Patients with more than 2nd and 3rd degree cystocele

Exclusion Criteria:

* Having endometriosis
* Having a history and/ or active pelvic inflammatory disease
* Having uterine fibroids
* Having an adnexal cyst with risk of malignancy
* Being pregnant

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of pelvic organ prolapsus in patients undergone lateral suspension performed via V-Notes | 6 months
  Assessment of pop-q quantification staging system before and 6 months after lateral suspension performed via V-notes
Incidence of pelvic organ prolapse/urinary Incontinence and sexual function in patients undergone lateral suspension performed via V-Notes | 6 months
  Assessment of pisq-12 Questionnaire in patients undergone lateral suspension performed via V-Notes

CONTACTS AND LOCATIONS:
Locations (1):
- Saglık Bilimleri University Istanbul Gaziosmanpa Trainig and Research Hospital, Istanbul, Turkey (Türkiye)